CLINICAL TRIAL: NCT04000308
Title: Quadratus Lumborum Block Type 2 Versus Wound Infiltration in Cesarean Section: a Randomized Controlled Trial
Brief Title: QLB vs. Wound Infiltration in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Lucovnik, assistant professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0120-251/2019/4
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Analgesia; Cesarean Section
Keywords: Analgesia; Cesarean Section; Quadratus Lumborum Block type 2; Wound Infiltration
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed in a 1:1 ratio using a computer generated randomization sequence. A sealed opaque envelope containing the study number will opened by an anesthetist nurse who will not be involved in the study. This anesthetist nurse will prepare the study medication and label the syringes with a unique study number which will be used to identify the study medication and will be revealed only on completion of data collection at the end of the study. The anesthetists, obstetricians, nurses who will be involved in the study, parturients, and other healthcare providers who will be involved in postoperative care will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block type 2 (Experimental): The obstetrician (multiple, experienced clinicians) will infiltrate the wound (Pfannenstiel incision) subcutaneously at the end of surgery with 20 ml normal saline. Subsequently, a US-guided QLB using a linear/convex transducer will be performed by the anesthesiologist using 30 ml levobupivacaine 0.18% (20 ml 0.25% levobupivacaine + 10 ml normal saline) bilaterally (60 ml in total).
  Interventions: Drug: Quadratus Lumborum Block type 2
- Wound Infiltration (Active Comparator): Patricipants will receive 20 ml levobupivacaine 0.25% infiltration in the surgical wound and US-guided QLB with 30 ml normal saline bilaterally (60 ml in total).
  Interventions: Drug: Wound Infiltration

INTERVENTIONS:
Drug: Quadratus Lumborum Block type 2 — The obstetrician (multiple, experienced clinicians) will infiltrate the wound (Pfannenstiel incision) subcutaneously at the end of surgery with 20 ml normal saline. Subsequently, a US-guided QLB using a linear/convex transducer will be performed by the anesthesiologist using 30 ml levobupivacaine 0.18% (20 ml 0.25% levobupivacaine + 10 ml normal saline) bilaterally (60 ml in total).
  Arms: Quadratus Lumborum Block type 2
Drug: Wound Infiltration — Participants will receive 20 ml levobupivacaine 0.25% infiltration in the surgical wound and US-guided QLB with 30 ml normal saline bilaterally (60 ml in total).
  Arms: Wound Infiltration

SUMMARY:
Effective postoperative analgesia after cesarean section (CS) is important because it enables early ambulation and facilitates breast-feeding. A 2009 Cochrane review concluded that wound infiltration with local analgesic after CS reduced opioid consumption. In addition, two regional anesthetic techniques, the transversus abdominis plane (TAP) block and the quadratus lumborum block (QLB), have been shown in multiple studies to reduce post-operative opioid consumption after CS. A recent randomized controlled trial showed that QLB is more effective in reducing morphine consumption post-CS compared to TAP. No randomized controlled trial to date, however, compared the analgesic effect of QLB with infiltration of the wound after CS. The objective of the study is to compare the analgesic effect of QLB type 2 with wound infiltration after CS.

DETAILED DESCRIPTION:
Effective postoperative analgesia after cesarean section (CS) is important because it enables early ambulation and facilitates breast-feeding. Post-CS analgesia is usually multimodal. At our hospital, patients are routinely given a combination of parenteral paracetamol, metamizole and tramadol at fixed intervals with additional intravenous piritramide on demand. The well-known side effects of piritramide (nausea, vomiting, and sedation) may interfere with interaction between mother and child, breast-feeding and post-partum experience in a dose-dependent manner. Alternative strategies to reduce rescue opioid analgesic consumption post-CS section are, therefore, required.

A 2009 Cochrane review concluded that wound infiltration with local analgesic after CS reduced opioid consumption. In addition, two regional anesthetic techniques, the transversus abdominis plane (TAP) block and the quadratus lumborum block (QLB), have been shown in multiple studies to reduce post-operative opioid consumption after CS. A recent randomized controlled trial showed that QLB is more effective in reducing morphine consumption post-CS compared to TAP.

Telnes et al. compared TAP block with wound infiltration with local anesthetic following CS. They found no reduction in cumulative morphine consumption and more pronounced sedation associated with TAP block. No randomized controlled trial to date, however, compared the analgesic effect of QLB with infiltration of the wound after CS.

The objective of the study is to compare the analgesic effect of QLB type 2 with wound infiltration after CS.

ELIGIBILITY:
Inclusion Criteria:

* Parturients scheduled for an elective caesarean delivery under spinal anaesthesia with an American Society of Anesthesiologists physical status I or II, singleton pregnancy, and gestational age ≥ 37 completed weeks.

Exclusion Criteria:

* Congenital or acquired coagulopathy.
* Allergy to local anaesthetics.
* History of drug abuse.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Total amount of piritramide used in first 24 hours | 24 hours post CS
  Total amount of piritramide administered in the first 24 hours after CS

SECONDARY OUTCOMES:
Total amount of piritramide used in first 48 hours | 48 hours post CS
  Total amount of piritramide administered in the first 48 hours after CS
Numerical rating scale (0-10) at rest | Within 48 hours post CS
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Numerical rating scale (0-10) with movement | Within 48 hours post CS
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Ramsay scale | within 24 hours post CS
  Ramsay scale measures level of sedation: 1 Patient is anxious and agitated or restless, or both. 2 Patient is co-operative, oriented, and tranquil. 3 Patient responds to commands only. 4 Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
Itching | within 24 hours post CS
  Itching will be assessed as following: 0, none; 1, mild; 2, moderate; and 3, severe
Nausea | within 24 hours post CS
  Nausea will be assessed as following: 0, none; 1, mild; 2, moderate; and 3, severe or vomiting
Surgery-to-first-ambulation time | within 48 hours post CS
  Time from surgery to first ambulation of the patient
Surgery-to-breast-feeding time | within 48 hours post CS
  Time from surgery to first breast-feeding

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stopar-Pintaric T, Blajic I, Visic U, Znider M, Plesnicar A, Vlassakov K, Lucovnik M. Posteromedial quadratus lumborum block versus wound infiltration after caesarean section: A randomised, double-blind, controlled study. Eur J Anaesthesiol. 2021 Aug 1;38(Suppl 2):S138-S144. doi: 10.1097/EJA.0000000000001531. PMID 33988528